CLINICAL TRIAL: NCT00770887
Title: Self Administration of Subcutaneous Depot Medroxyprogesterone Acetate: A Pilot Observational Study of Feasibility and Acceptability
Brief Title: Self Administration of Subcutaneous Depot Medroxyprogesterone Acetate
Acronym: SAD
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Pfizer (Industry); Planned Parenthood Federation of America (Other)
Responsible Party: Sujatha Prabhakaran MD, MPH Medical Director, Planned Parenthood of Southwest and Central Florida
Other Study IDs: 08-2404
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Fertility
Keywords: Undesired fertility
MeSH Terms: interventions — Self Administration

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study participants: This study will enroll 50 English-speaking/literate women at least 18 years of age of any race who have sought contraception with DMPA at the Planned Parenthood of Southwest and Central Florida clinics in Tampa and Fort Myers. Patients who choose to begin DMPA or who have already been using DMPA will be approached regarding voluntary participation in the study. Because DMPA is contraindicated in pregnancy, women with a positive urine pregnancy will not be eligible. Should a woman become pregnant during the study, she will receive no further DMPA injections
  Interventions: Procedure: Self administration

INTERVENTIONS:
Procedure: Self administration — Subjects will self administer injections of 104 mg of the subcutaneous formulation of depot medroxyprogesterone acetate (depo-subQ provera 104).

SUMMARY:
The purpose of this study is to assess continuation rates and patient satisfaction with self administration subcutaneous depot medroxyprogesterone acetate.

DETAILED DESCRIPTION:
This observational study will include new or current Depo Provera users who express interest in attempting subcutaneous self administration of depot medroxyprogesterone acetate. Candidates will be taught self administration by a clinic assistant at Planned Parenthood of Southwest and Central Florida. Patients who are able to correctly self administer the medication and wish to attempt to continue home self administration, will be provided the supplies and educational materials to do so. Continuation rates and satisfaction with this method will be assessed using preaddressed surveys that patients will return with the above information.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older
* Can understand written and spoken English
* Current or past user of DMPA or desires initiation of DMPA for contraception
* Provider has approved DMPA use in this woman
* Willing to consider/attempt DMPA self-injection.
* Willing to receive phone calls/letter for follow up
* Willing to return letters for follow up

Exclusion Criteria:

Has contraindications to DMPA use:

* Vaginal bleeding of unknown etiology
* Medication use for Cushing's syndrome
* Currently pregnant
* Blood pressure >160/100
* Intolerance to the idea of irregular or absent menses

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will enroll 50 English-speaking/literate women at least 18 years of age of any race who have sought contraception with DMPA at the Planned Parenthood of Southwest and Central Florida in Tampa and Fort Myers. Patients who choose to begin DMPA or who have already been using DMPA will be approached regarding voluntary participation in the study. Because DMPA is contraindicated in pregnancy, women with a positive urine pregnancy will not be eligible. Should a woman become pregnant during the study, she will receive no further DMPA injections
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with/feasibility of self injection of subcutaneous depot medroxyprogesterone acetate | At onset of trial and every 12 weeks for 1 year

SECONDARY OUTCOMES:
Continuation rates of depot medroxyprogesterone acetate among self-injectors | Every 12 weeks for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sujatha Prabhakaran, MD, Principal Investigator — Planned Parenthood of Southwest and Central Florida
Locations (2):
- United States (2):
  - Planned Parenthood of Southwest and Central Florida, Fort Myers, Florida
  - Planned Parenthood of Southwest and Central Florida, Tampa, Florida

REFERENCES:
- [Background] Potter LS, Dalberth BT, Canamar R, Betz M. Depot medroxyprogesterone acetate pioneers. A retrospective study at a North Carolina Health Department. Contraception. 1997 Nov;56(5):305-12. doi: 10.1016/s0010-7824(97)00160-1. PMID 9437559
- [Background] Nelson AL, Katz T. Initiation and continuation rates seen in 2-year experience with Same Day injections of DMPA. Contraception. 2007 Feb;75(2):84-7. doi: 10.1016/j.contraception.2006.09.007. Epub 2006 Oct 31. PMID 17241834
- [Background] Rickert VI, Tiezzi L, Lipshutz J, Leon J, Vaughan RD, Westhoff C. Depo Now: preventing unintended pregnancies among adolescents and young adults. J Adolesc Health. 2007 Jan;40(1):22-8. doi: 10.1016/j.jadohealth.2006.10.018. PMID 17185202
- [Background] Moreau C, Cleland K, Trussell J. Contraceptive discontinuation attributed to method dissatisfaction in the United States. Contraception. 2007 Oct;76(4):267-72. doi: 10.1016/j.contraception.2007.06.008. Epub 2007 Aug 28. PMID 17900435
- [Background] Lim SW, Rieder J, Coupey SM, Bijur PE. Depot medroxyprogesterone acetate use in inner-city, minority adolescents: continuation rates and characteristics of long-term users. Arch Pediatr Adolesc Med. 1999 Oct;153(10):1068-72. doi: 10.1001/archpedi.153.10.1068. PMID 10520615
- [Background] Drug Information. [Internet]. Rockville, MD: United States Food and Drug Administration; CDER Drug and Biologic Approvals for Calendar Year 2004; [cited December 12, 2007]. Available from: http://www.fda.gov/cder/rdmt/ndaaps04cy.htm
- [Background] Jain J, Jakimiuk AJ, Bode FR, Ross D, Kaunitz AM. Contraceptive efficacy and safety of DMPA-SC. Contraception. 2004 Oct;70(4):269-75. doi: 10.1016/j.contraception.2004.06.011. PMID 15451329
- [Background] Rodger MA, King L. Drawing up and administering intramuscular injections: a review of the literature. J Adv Nurs. 2000 Mar;31(3):574-82. doi: 10.1046/j.1365-2648.2000.01312.x. PMID 10718876
- [Background] Watts AC, Howie CR, Simpson AH. Assessment of a self-administration protocol for extended subcutaneous thromboprophylaxis in lower limb arthroplasty. J Bone Joint Surg Br. 2006 Jan;88(1):107-10. doi: 10.1302/0301-620X.88B1.17003. PMID 16365131
- [Background] Nichols J, Knochenhauer E, Fein SH, Nardi RV, Marshall DC. Subcutaneously administered Repronex in oligoovulatory female patients undergoing ovulation induction is as effective and well tolerated as intramuscular human menopausal gonadotropin treatment. Fertil Steril. 2001 Jul;76(1):58-66. doi: 10.1016/s0015-0282(01)01856-8. PMID 11438320
- [Background] Becker WJ, Riess CM, Hoag J. Effectiveness of subcutaneous dihydroergotamine by home injection for migraine. Headache. 1996 Mar;36(3):144-8. doi: 10.1046/j.1526-4610.1996.3603144.x. PMID 8984085
- [Background] Stanwood NL, Eastwood K, Carletta A. Self-injection of monthly combined hormonal contraceptive. Contraception. 2006 Jan;73(1):53-5. doi: 10.1016/j.contraception.2005.05.020. Epub 2005 Nov 14. PMID 16371295
- [Background] Bahamondes L, Marchi NM, Nakagava HM, de Melo ML, Cristofoletti Mde L, Pellini E, Scozzafave RH, Petta C. Self-administration with UniJect of the once-a-month injectable contraceptive Cyclofem. Contraception. 1997 Nov;56(5):301-4. doi: 10.1016/s0010-7824(97)00162-5. PMID 9437558
- [Background] Lakha F, Henderson C, Glasier A. The acceptability of self-administration of subcutaneous Depo-Provera. Contraception. 2005 Jul;72(1):14-8. doi: 10.1016/j.contraception.2004.12.002. PMID 15964286
- [Background] Mosher WD, Martinez GM, Chandra A, Abma JC, Willson SJ. Use of contraception and use of family planning services in the United States: 1982-2002. Adv Data. 2004 Dec 10;(350):1-36. PMID 15633582